CLINICAL TRIAL: NCT02796547
Title: Randomized Double Blind Clinical Trial on the Effect of Levobupivacaine Infiltration Versus Placebo on the Post Partum Perineal Pain in Episiotomy in Primiparous Women After Instrumental Delivery
Brief Title: Effect of Levobupivacaine Infiltration on the Post Partum Perineal Pain in Episiotomy, in Primiparous Women After Instrumental Delivery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of human ressources
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUB-EQUIDOL
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Episiotomy
Keywords: Episiotomy; Levobupivacaine
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine (Experimental): Primiparous patients in whom a instrumental delivery with episiotomy is conducted. The infiltration of the banks of the episiotomy will be done with Levobupivacaine. This is the only intervention specific to the study, as compared to the standard of care.
  Interventions: Drug: Levobupivacaine
- Placebo (Placebo Comparator): Primiparous patients in whom a instrumental delivery with episiotomy is conducted. The infiltration of the banks of the episiotomy will be done with physiological serum.This is the only intervention specific to the study, as compared to the standard of care.
  Interventions: Other: Physiological serum

INTERVENTIONS:
Drug: Levobupivacaine — Infiltration of the banks of the episiotomy done with Levobupivacaine
  Arms: Levobupivacaine
Other: Physiological serum — Infiltration of the banks of the episiotomy done with physiological serum
  Arms: Placebo

SUMMARY:
An episiotomy is an incision of the perineum to facilitate childbirth by natural means. Perineal pain are more frequent and intense if the incision of the perineum is important. In particular, simple vaginal or perineal tears are less painful than episiotomies in the first seven days postpartum, whereas at six weeks postpartum, there is no significant difference anymore.The patients are the most symptomatic in the immediate postnatal period, but the pain may persist up to 2 weeks after delivery in 20 to 25% of cases. These pains are often undervalued and may interfere with the mother-child bond in the absence of an effective treatment. Perineal pain are usually treated with painkillers, in particular non-steroidal anti-inflammatory drugs given orally or rectally and paracetamol.

The scar infiltration is one of the components of a multimodal postoperative analgesia strategy. It consists in the simultaneous use of several drugs or analgesic techniques, acting on different pain components in order to improve the overall efficiency.The most used local anesthetics at present are bupivacaine, ropivacaine and levobupivacaine.Ropivacaine has a lesser vasodilatory effect than bupivacaine, resulting in longer persistence at the injection point and a blood resorption that is more spread. The systemic toxicity threshold is also higher. Levobupivacaine is the enantiomer of bupivacaine. It has vascular effects, and an intermediate systemic toxicity threshold intermediate between bupivacaine and ropivacaine. Lidocaine has a limited duration of action. Its use is interesting in complement infiltrations when a rapid onset of action is desired.

So far, there is no data in the literature regarding the effect of levobupivacaine in episiotomies associated pain. The objective of this study is to evaluate the effect of local injections of levobupivacaine on episiotomies associated pain.

DETAILED DESCRIPTION:
An episiotomy is an incision of the perineum to facilitate childbirth by natural means. This gesture is performed in 68% of primiparous women and 31% of multiparous women, according to Audipog data of 2003, with a downward trend since the 80's. The episiotomy reduces the risk of occurrence of anterior perineal tears, but has no preventive effect on 3rd and 4th grade perineal tears, according to the Anglo-Saxon classification. The French national college of obstetricians and gynecologists (CNGOF) recommends thus a restrictive use of episiotomy. Perineal pain are more frequent and intense if the incision of the perineum is important. In particular, simple vaginal or perineal tears are less painful than episiotomies in the first seven days postpartum, whereas at six weeks postpartum, there is no significant difference anymore.The patients are the most symptomatic in the immediate postnatal period, but the pain may persist up to 2 weeks after delivery in 20 to 25% of cases. These pains are often undervalued and may interfere with the mother-child bond in the absence of an effective treatment. Perineal pain are usually treated with painkillers, in particular non-steroidal anti-inflammatory drugs given orally or rectally and paracetamol.

The scar infiltration is one of the components of a multimodal postoperative analgesia strategy. It consists in the simultaneous use of several drugs or analgesic techniques, acting on different pain components in order to improve the overall efficiency. This also reduces the consumption of analgesics having multiple side effects, such as opioids. Local anesthetics act at several levels. First, they block the transmission of pain messages at the nocireceptors level and have an analgesic effect on the nearby surgery site. The immediate post-operative pain is thus diminished. Furthermore, by blocking the pain message at the peripheric level, local anesthetics might have an effect on the formation of central hyperalgesia, responsible for longer-term pain. The local anesthetics also have local and systemic anti-inflammatory properties, that may have an effect on postoperative pain and on the establishment of hyperalgesic phenomena.

The most used local anesthetics at present are bupivacaine, ropivacaine and levobupivacaine. Ropivacaine has a lesser vasodilatory effect than bupivacaine, resulting in longer persistence at the injection point and a blood resorption that is more spread. The systemic toxicity threshold is also higher. Levobupivacaine is the enantiomer of bupivacaine. It has vascular effects, and an intermediate systemic toxicity threshold intermediate between bupivacaine and ropivacaine. Lidocaine has a limited duration of action. Its use is interesting in complement infiltrations when a rapid onset of action is desired.

Many scar infiltration indications are documented in the literature, such as inguinal hernias, hemorrhoids cures, thyroidectomy, orthopedic surgery, breast surgery, and cesarean section.Various studies evaluated the effectiveness of different local anesthetics in episiotomies and perineal tears.

So far, there is no data in the literature regarding the effect of levobupivacaine in episiotomies associated pain. The objective of this study is to evaluate the effect of local injections of levobupivacaine on episiotomies associated pain.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* Vaginal delivery with instrumentation (Suzor forceps, vacuum extraction, Thierry spatulas) with episiotomy
* Fœtus In cephalic position
* Single pregnancy
* Patient at least 18 years old
* Term superior or equal to 37 weeks of amenorrhea
* Patient under epidural analgesia
* Patient affiliated to a social security scheme
* Good understanding of French

Exclusion Criteria:

* Ineffective epidural analgesia, defined by the need for additional local anesthesia for episiotomy repair
* Perineal tear of the 3rd or 4th grade, according to the Anglo-Saxon classification
* Contra indications to levobupivacaine, paracetamol, ketoprofen
* Participation refusal
* Postpartum hemorrhage requiring arterial embolization, reoperation (evacuation of a vaginal thrombus, vessel ligation, hysterectomy by laparotomy) or placement of a Bakri® balloon.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
ENS pain scale | 24h post partum
  Pain evaluation on a simple numeric scale (ENS)

SECONDARY OUTCOMES:
Painkillers (ketoprofen) quantity | During the first 48h post partum
  Cumulated quantity of painkillers taken in addition to paracetamol in the first 48h post partum. Painkillers are given according to standard of care and are not a intervention specific to the study.
Painkillers (nefopam) quantity | During the first 48h post partum
  Cumulated quantity of painkillers taken in addition to paracetamol in the first 48h post partum.Painkillers are given according to standard of care and are not a intervention specific to the study.
Painkillers (ketoprofen) quantity | At day 15 post-partum
  Quantity of painkillers taken at day 15 post-partum. Painkillers are given according to standard of care and are not a intervention specific to the study.
Painkillers (nefopam) quantity | At day 15 post-partum
  Quantity of painkillers taken at day 15 post-partum. Painkillers are given according to standard of care and are not a intervention specific to the study.
Painkillers (paracetamol) quantity | At day 15 post-partum
  Quantity of painkillers taken at day 15 post-partum. Painkillers are given according to standard of care and are not a intervention specific to the study.
ENS pain scale | At day 15 post-partum
  Pain evaluation on a simple numeric scale (ENS)
Presence/absence of complications | At day 15 post-partum
  The quality of cicatrisation of the episiotomy will be assessed in order to track complications.
Likert scale | Day 1 post partum
  Impact of pain secondary to episiotomy on the activities of daily life (sitting, walking, urination, sleep, child care), assessed by the Likert scale
Likert scale | Day 2 post partum
  Impact of pain secondary to episiotomy on the activities of daily life (sitting, walking, urination, sleep, child care), assessed by the Likert scale
Likert scale | Day 15 post partum
  Impact of pain secondary to episiotomy on the activities of daily life (sitting, walking, urination, sleep, child care), assessed by the Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann; Florent FUCHS, MD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- CHU Brugmann, Brussels, Belgium
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Background] Vendittelli F, Gallot D. [What are the epidemiologic data in regard to episiotomy?]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S12-1S23. French. PMID 16495823
- [Background] de Tayrac R, Panel L, Masson G, Mares P. [Episiotomy and prevention of perineal and pelvic floor injuries]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S24-1S31. French. PMID 16495824
- [Background] College National de Gynecolegues et Obstetriciens Francais. [Text of the guideline for episiotomy]. J Gynecol Obstet Biol Reprod (Paris). 2006 Feb;35(1 Suppl):1S77-1S80. No abstract available. French. PMID 16495830
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Albers L, Garcia J, Renfrew M, McCandlish R, Elbourne D. Distribution of genital tract trauma in childbirth and related postnatal pain. Birth. 1999 Mar;26(1):11-7. doi: 10.1046/j.1523-536x.1999.00011.x. PMID 10352050
- [Background] Peter EA, Janssen PA, Grange CS, Douglas MJ. Ibuprofen versus acetaminophen with codeine for the relief of perineal pain after childbirth: a randomized controlled trial. CMAJ. 2001 Oct 30;165(9):1203-9. PMID 11706909
- [Background] Hedayati H, Parsons J, Crowther CA. Rectal analgesia for pain from perineal trauma following childbirth. Cochrane Database Syst Rev. 2003;(3):CD003931. doi: 10.1002/14651858.CD003931. PMID 12917995
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Marret E, Kurdi O, Zufferey P, Bonnet F. Effects of nonsteroidal antiinflammatory drugs on patient-controlled analgesia morphine side effects: meta-analysis of randomized controlled trials. Anesthesiology. 2005 Jun;102(6):1249-60. doi: 10.1097/00000542-200506000-00027. PMID 15915040
- [Background] Brennan TJ, Zahn PK, Pogatzki-Zahn EM. Mechanisms of incisional pain. Anesthesiol Clin North Am. 2005 Mar;23(1):1-20. doi: 10.1016/j.atc.2004.11.009. PMID 15763408
- [Background] Kawamata M, Watanabe H, Nishikawa K, Takahashi T, Kozuka Y, Kawamata T, Omote K, Namiki A. Different mechanisms of development and maintenance of experimental incision-induced hyperalgesia in human skin. Anesthesiology. 2002 Sep;97(3):550-9. doi: 10.1097/00000542-200209000-00006. PMID 12218519
- [Background] Sanford M, Keating GM. Levobupivacaine: a review of its use in regional anaesthesia and pain management. Drugs. 2010 Apr 16;70(6):761-91. doi: 10.2165/11203250-000000000-00000. PMID 20394458
- [Background] Ausems ME, Hulsewe KW, Hooymans PM, Hoofwijk AG. Postoperative analgesia requirements at home after inguinal hernia repair: effects of wound infiltration on postoperative pain. Anaesthesia. 2007 Apr;62(4):325-31. doi: 10.1111/j.1365-2044.2007.04991.x. PMID 17381566
- [Background] Franchi M, Cromi A, Scarperi S, Gaudino F, Siesto G, Ghezzi F. Comparison between lidocaine-prilocaine cream (EMLA) and mepivacaine infiltration for pain relief during perineal repair after childbirth: a randomized trial. Am J Obstet Gynecol. 2009 Aug;201(2):186.e1-5. doi: 10.1016/j.ajog.2009.04.023. Epub 2009 Jun 26. PMID 19560111
- [Background] Minassian VA, Jazayeri A, Prien SD, Timmons RL, Stumbo K. Randomized trial of lidocaine ointment versus placebo for the treatment of postpartum perineal pain. Obstet Gynecol. 2002 Dec;100(6):1239-43. doi: 10.1016/s0029-7844(02)02339-6. PMID 12468168
- [Background] Kafali H, Iltemur Duvan C, Gozdemir E, Simavli S, Ozturk Turhan N. Placement of bupivacaine-soaked Spongostan in episiotomy bed is effective treatment modality for episiotomy-associated pain. J Minim Invasive Gynecol. 2008 Nov-Dec;15(6):719-22. doi: 10.1016/j.jmig.2008.08.006. PMID 18971135
- [Background] Sillou S, Carbonnel M, N'Doko S, Dhonneur G, Uzan M, Poncelet C. [Postpartum perineal pain: effectiveness of local ropivacaine infiltration]. J Gynecol Obstet Biol Reprod (Paris). 2009 Oct;38(6):510-5. doi: 10.1016/j.jgyn.2009.03.008. Epub 2009 Jun 2. French. PMID 19493636